CLINICAL TRIAL: NCT00505661
Title: Phase II Study of Letrozole in Patients With Recurrent Advanced Borderline Tumors or Low Grade Epithelial Cancers of the Ovary, Fallopian Tube and Primary Peritoneum
Brief Title: Letrozole in Patients With Ovarian Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow patient accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0486
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Letrozole; Femara
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole (Experimental): 2.5 mg by mouth (PO) daily
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — 2.5 mg PO Once Daily
  Other Names: Femara

SUMMARY:
Primary Objectives:

* To determine the objective response rate of Letrozole when administered to patients with advanced or recurrent borderline tumors or low-grade epithelial cancers from the ovary , fallopian tube or peritoneum.
* To determine the time to tumor progression of patients with advanced or recurrent borderline tumors or low-grade epithelial cancers from the ovary, fallopian tube or peritoneum.
* To identify the biological markers to predict response to Letrozole and study the aspects of the hormones in these types of tumors.

DETAILED DESCRIPTION:
Letrozole is an anticancer hormone that is FDA approved for use in patients with advanced breast cancer.

Before you can be enrolled in this study, you must go through some screening tests to make sure you are eligible. The screening tests include a complete medical history and physical exam, including measurement of your pulse rate, breathing rate, temperature, height, weight, and blood pressure. The physical examination will also include measurement of any visible cancer lesions. You will be asked what medications you are taking, including over the counter medications, herbal medications, and vitamins. You will have chest x-rays and/or CT or MRI scans to measure the size of your tumors. You will have routine blood tests (about 2 and a 1/2 tablespoons) performed.

If you qualify for the study, you will take Letrozole once a day by mouth. Letrozole will be dispensed in the form of a tablet. Four to eight weeks worth of Letrozole will be prescribed to you by your treatment doctor at each visit. You will continue to receive Letrozole as long as you are responding to treatment.

You will be required to come back for check-up at least once every 2 months while on study for the first two years. You should contact the study doctor if you feel unwell or feel the need to see the doctor before your appointment earlier than your designated appointment.

At each follow-up visit, you will have a complete physical exam. The chest x-rays and/or CT or MRI scans will be repeated every 2 months, and at the time you complete the trial, or at any other time if necessary. Blood tests (about 1 tablespoon) will be performed every 2 months. Information about the medications you are taking, or medical problems you have had since your last visit will be collected. At each follow-up visit, you will also be asked to complete a one page, paper and pencil check off sheet. You will be asked to identify symptoms you may be having and to note the amount of distress each symptom is causing you.

You will be taken off study if the disease gets worse or intolerable side effects occur and your doctor will discuss possible treatment options with you.

However, as long as you continue to benefit from Letrozole treatment, you will continue on this treatment. If you are on letrozole treatment beyond two years, you will be followed up at three months interval. At these follow up visits, you will be asked questions about your medical history and have a physical exam. You will also have blood (about tablespoon) and urine tests, and/or radiological evaluation of the tumor. As long as you continue to benefit from letrozole treatment, you will be followed up.

Your status will be followed for as long as possible even after you are taken off the study drug. You will be contacted by phone or asked to come to the clinic for a routine visit. You will be contacted every 6 weeks for 1 year after the study and every 12 weeks for the rest of your life.

This is an investigational study. Letrozole is not approved by the FDA for the treatment of recurrent low grade or borderline ovarian, fallopian tube or primary peritoneal cancer. A total of up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. History of histologically confirmed diagnosis of borderline tumors or low-grade epithelial cancer from the ovary, fallopian tube or primary peritoneum. Eligible histologies include borderline serous papillary, borderline mucinous papillary, borderline endometrioid, low-grade serous papillary, low-grade mucinous papillary, low-grade endometrioid and mixture of the above. Patients whose tumors are histologically borderline but have low grade invasive implants are also included. Patients whose tumors are histologically borderline but which include high grade components are excluded.
2. Recurrent or advanced borderline or low-grade epithelial ovarian, fallopian tube or primary peritoneal tumors not amenable to surgery, or patients who have measurable residual disease at the end of secondary cytoreduction.
3. The ovarian tumors have to be either estrogen receptor or progesterone receptor positive.
4. Measurable disease by radiological imaging studies. Raised CA125 tumor marker alone and lesions located in previously irradiated areas are not considered measurable.
5. Age greater than 18 years of age.
6. Expected survival of more than 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
8. Willingness to comply with study procedures and follow up examinations.
9. Have written informed consent. (Signature on consent form indicating that the patient is aware of the nature of her disease and willingly gives written consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternative treatment options and potential benefits and risks associated with the therapy).
10. Known history of Central nervous system metastases allowed if patients have had treatment, are neurologically stable, and do not require oral or intravenous steroids or anti-convulsants, provided brain scan (Computer Assisted Tomography or Magnetic Resonance Imaging Scans) shows absence of active disease.
11. Have adequate bone marrow reserve as indicated by absolute neutrophil count (ANC)> 1,500/ mm3; platelet count > 100,000/mm3; hemoglobin > 9.0g/dL.
12. Have adequate liver function tests as indicated by bilirubin < 1.5 X normal, alanine amino-transferase (ALT)< 3 X normal; and aspartate amino-transferase (AST) < 3 X normal.
13. Have adequate renal function tests as indicated by serum creatinine of < 1.5mg/dl.

Exclusion Criteria:

1. Failure to recover from any prior surgery or major surgery within 4 weeks of study entry
2. Patients with sarcomatous, germ cell or stromal elements in their cancers are not eligible.
3. Patients with intermediate and high-grade primary ovarian, fallopian tube, and primary peritoneal epithelial carcinoma. Patients whose tumors are histologically borderline but which includes high grade components are excluded.
4. Pregnant or lactating women
5. Leptomeningeal or carcinomatous meningitis
6. Unstable medical conditions such as uncontrolled cardiac arrythmia or history of myocardial infarction within 6 months
7. Any severe, concurrent disease, infection or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for study entry.
8. Any signs of intestinal obstruction interfering with nutrition
9. Treatment with chemotherapy, radiotherapy, radiopharmaceuticals or immunotherapy within 4 weeks of first study dosing with letrozole (within 6 weeks for nitrosureas or mitomycin C) or failure to recover from the toxic effects of any of these therapies prior to study entry.
10. Patients with more than 4 prior chemotherapy regimes with all platinum regimes counted as one.
11. Patients who has had prior anti-cancer hormonal therapy for ovarian cancer with aromatase inhibitors. Patients treated with gonadotrophin agonist, gonadotropin antagonist and Selective estrogen receptor modulators (SERMS) are allowed. Patients on hormone replacement therapy or who have had fertility treatment with estrogens and gonadotropins are also allowed.
12. Patients on estrogen and progesterone replacement therapy must have a wash out period of 4 weeks.
13. A history of prior malignancy except for adequately treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, or other cancer for which the patient has not been disease- free for at least five years
14. Patients receiving concurrent chemotherapy, radiotherapy or immunotherapy.
15. Participation in any investigational drug study within 30 days of the first day of dosing.
16. Psychiatric disorders that would preclude obtaining informed consent and participation in an ongoing research study
17. Patients with a known history of human immunodeficiency virus (HIV) infection
18. Patients with inadequately treated serious thromboembolic disease such as pulmonary embolism and deep vein thrombosis, or with known clotting disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Kavanagh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 09/24/03 through 01/30/08. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to slow patient accrual.
Period: Overall Study
Arm/Group | Letrozole
Started | 16
Completed | 12
Not Completed | 4
Not completed — Not Eligible | 4

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole
Number analyzed (Participants) | 16
Age Continuous [Median (Full Range); unit: years] | 54 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Following Treatment With Letrozole
Description: Using RECIST criteria, Objective Response evaluated every 2 months.
Time Frame: 2 month intervals for first 2 years
Population: Analysis was per protocol, only 9 of 12 eligible patients were evaluable for response.
Measure: Number; unit: participants
Arm/Group | Letrozole
Number analyzed (Participants) | 9
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 6

ADVERSE EVENTS:
Time Frame: 4 years and 4 months
Arm/Group | Letrozole
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=16)
Fatigue (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No